CLINICAL TRIAL: NCT07346391
Title: Clinical Effectiveness of Combining Free Gingival Strip Graft With Platelet-Rich Fibrin for Peri-Implant Keratinized Mucosa Augmentation
Brief Title: Augmentation of Peri-implant Keratinized Mucosa Using a Combination of Free Gingival Graft Strip With Platelet-Rich Fibrin
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nguyen Van Khuong (Other)
Responsible Party: Sponsor-Investigator, Nguyen Van Khuong, Doctor, University of Medicine and Pharmacy at Ho Chi Minh City
Organization: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25309-DHYD
Record Dates: First submitted 2025-12-23; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Dental Implants
Keywords: Combination technique of strip free gingival grafts and PRF in augmenting keratinized mucosa around dental implants
MeSH Terms: interventions — Prolactin-Releasing Hormone; fibrinopeptides gamma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The soft tissue aesthetic outcomes are evaluated by an independent assessor who is blinded to the treatment groups (the assessor does not know which group the patient being evaluated belongs to).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Free Gingival Graft (FGG) (Experimental): A surgical procedure where a graft consisting of epithelium and connective tissue is harvested from the palate and transplanted to the peri-implant area to increase the width and height of keratinized mucosa
  Interventions: Procedure: Conventional Free Gingival Graft (FGG) to increase keratinized mucosa around dental implants
- Combining a strip free gingival graft with Platelet-Rich Fibrin (PRF) to increase keratinized mucosa (Experimental): Venous blood is collected using a butterfly needle and 10ml tubes to prepare the PRF membrane. A keratinized mucosa strip of appropriate dimensions is harvested from the patient's palate. The strip free gingival graft and PRF membrane are then sutured and stabilized at the recipient site.
  Interventions: Procedure: Combining a strip free gingival graft (sFGG) with Platelet-Rich Fibrin (PRF) to increase keratinized mucosa around dental implants

INTERVENTIONS:
Procedure: Combining a strip free gingival graft (sFGG) with Platelet-Rich Fibrin (PRF) to increase keratinized mucosa around dental implants — Venous blood is collected using a butterfly needle and 10ml tubes to prepare the PRF membrane. A keratinized mucosa strip of appropriate dimensions is harvested from the patient's palate. The strip free gingival graft and PRF membrane are then sutured and stabilized at the recipient site.
  Arms: Combining a strip free gingival graft with Platelet-Rich Fibrin (PRF) to increase keratinized mucosa
Procedure: Conventional Free Gingival Graft (FGG) to increase keratinized mucosa around dental implants — A surgical procedure where a graft consisting of epithelium and connective tissue is harvested from the palate and transplanted to the peri-implant area to increase the width and height of keratinized
  Arms: Conventional Free Gingival Graft (FGG)

SUMMARY:
This clinical trial aims to evaluate the clinical effectiveness of combining a strip free gingival graft (sFGG) with Platelet-Rich Fibrin (PRF) for increasing keratinized mucosa around dental implants. The study compares this combined technique with the conventional free gingival graft (FGG) method through three primary objectives:

1. comparing the increase in keratinized mucosal height at immediate post-op, 1, 4, and 6 months;
2. assessing post-operative pain levels at 1, 3, 7, and 14 days;
3. evaluating soft tissue aesthetic outcomes at 4 and 6 months post-surgery.

DETAILED DESCRIPTION:
Pre-operative phase:

Eligible patients undergo clinical examination and medical record documentation. Written informed consent is obtained prior to enrollment. Participants are randomly assigned by drawing one of 22 sealed envelopes: odd numbers are allocated to Group A (strip free gingival graft with PRF) and even numbers to Group B (conventional free gingival graft). Baseline intraoral and extraoral photographs and intraoral scans (PLY format) are obtained.

Intra-operative phase:

* Group A (Experimental): PRF is prepared from venous blood. A strip free gingival graft is harvested from the palate and placed at the recipient site in combination with PRF.
* Group B (Control): A conventional free gingival graft is harvested from the palate and placed at the recipient site.

Post-operative phase:

Follow-up visits are conducted at days 1, 3, 7, and 14, and at 1, 4, and 6 months post-surgery. At 1 month, healing abutments are placed and prosthetic treatment begins. Keratinized mucosa changes are assessed using pre- and post-operative intraoral scans. Post-operative pain is evaluated using the Visual Analog Scale (VAS), and soft tissue aesthetic outcomes are assessed at 4 and 6 months using a standardized aesthetic score.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting the following criteria are eligible for the study:

  * Prosthetic Phase: Patients scheduled for the prosthetic phase of dental implant treatment.
  * Keratinized Mucosa: Keratinized mucosa height (buccal or lingual) of less than 2 mm around the implant.
  * Systemic Health: Systemic health status classified as ASA I or II according to the American Society of Anesthesiologists classification.
  * Oral Hygiene: Good oral hygiene, defined by a mean full-mouth plaque index (PlI) of ≤ 1.

Exclusion Criteria:

* Patients meeting any of the following criteria will be excluded from the study:

  * Systemic Conditions: Presence of systemic diseases or use of medications known to affect the oral mucosa or gingival health.
  * Periodontal Health: Untreated periodontal disease and/or peri-implant diseases.
  * Surgical History: History of mucogingival surgery at the intended surgical site.
  * Pregnancy/Lactation: Pregnant or breastfeeding women.
  * Oral Hygiene: Poor oral hygiene, defined by a mean full-mouth plaque index (PlI) > 1.
  * Smoking: Current smokers.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-12-24 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of the increase in peri-implant keratinized mucosa width | 1, 4, 6 months
  KMW was assessed at the mid-buccal aspect of each implant, measuring the distance from the MGJ to the mucosal margin/alveolar zenith using STL surface data at 1, 4, and 6 months.
Soft tissue esthetics assessed by the modified Pink Esthetic Score (PES) | 4 months and 6 months post-operatively
  "The esthetic outcome of the peri-implant soft tissue is evaluated using the modified Pink Esthetic Score (PES) as described by Fürhauser et al. (2005). The assessment compares the grafted area to the adjacent natural tooth based on seven parameters: Soft tissue color difference, soft tissue texture difference, grafted site margins-mesial side, distal side, level of mucogingival junction, keloid-like appearance.
  Each parameter is assigned a score of 0, 1, or 2 (0 being the lowest, 2 being the highest/most esthetic). The total PES score ranges from 0 to 14, where a higher score indicates a superior esthetic result
Post-operative pain intensity measured by Visual Analog Scale (VAS) | 1, 3, 7 and 14 days post-operatively
  Pain intensity is measured on a Visual Analog Scale from 0 (no pain) to 10 (unbearable pain). Participants will be asked to mark their level of discomfort at each time point.